CLINICAL TRIAL: NCT03545789
Title: Phase 1 Test-retest Evaluation of [18F]MNI-958 PET as an Imaging Marker for Tau Protein in the Brain of Patients With Alzheimer's Disease and Probable PSP as Compared to Healthy Volunteers
Brief Title: Phase 1 Test-retest Evaluation of [18F]MNI-958 PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F]MNI-958 Test-Retest
Record Dates: First submitted 2018-03-15; First posted 2018-06-04 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers; Alzheimer Disease; Progressive Supranuclear Palsy
Keywords: HV; AD; PSP
MeSH Terms: conditions — Alzheimer Disease; Supranuclear Palsy, Progressive | interventions — florbetapir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]MNI-958 (Experimental): To measure blood metabolites of [18F]MNI-958 and perform kinetic modeling to assess its ability to measure tau protein in brain using the tracer plasma concentration or a reference region as indirect input.
  Interventions: Drug: [18F]MNI-958

INTERVENTIONS:
Drug: [18F]MNI-958 — Subjects will undergo PET imaging using [18F]MNI-958, a PET radioligand for imaging tau.
  Other Names: [18F]Florbetapir

SUMMARY:
The overall goal of this protocol is to evaluate [18F]MNI-958 also known as APN-0000455 or PM-PBB3, a tau targeted radiopharmaceutical.

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate [18F]MNI-958 also known as APN-0000455 or PM-PBB3, a tau targeted radiopharmaceutical. The specific objectives are:

* To measure the dynamic uptake and washout of [18F]MNI- 958 in brain using positron emission tomography (PET) in patients with Alzheimer's disease, Progressive Supranuclear Palsy and healthy volunteers.
* To measure blood metabolites of [18F]MNI-958 and perform kinetic modeling to assess its ability to measure tau protein in brain using the tracer plasma concentration or a reference region as indirect input.
* To obtain test/retest reliability of the tracer binding parameters in patients with Alzheimer's disease, Progressive Supranuclear Palsy and healthy volunteers.
* To acquire safety data following injection of [18F]MNI-958.

ELIGIBILITY:
Inclusion Criteria (for all subjects):

* Written informed consent must be obtained before any assessment is performed.
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of childbearing potential, must commit to use a barrier contraception method for the duration of the study.
* Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects for the study duration.
* Male subjects must not donate sperm for the study duration.
* Willing and able to cooperate with study procedures

Inclusion criteria for healthy volunteer subjects

* Males and females aged ≥50 years. Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the [18F]MNI-958 imaging visit.
* No cognitive impairment from neuropsychological battery as judged by the investigator
* Have screening or prior (in the last 90 days) amyloid PET imaging demonstrating no significant amyloid binding based on qualitative (visual read).
* No family history of Alzheimer's disease or neurological disease associated with dementia
* Have a CDR global score=0
* Have an MMSE score ≥28
* Willing and able to cooperate with study procedures

Inclusion criteria for subjects with a diagnosis of probable

Alzheimer's disease (AD):

* Males and females aged 50 to 80 years.
* Have probable Alzheimer's disease dementia, based on the NINCDS/ADRDA and DSM-IV criteria, with mild severity and amnestic presentation
* Have a CDR score ≥ 0.5 at screening
* Have a MMSE score between ≤ 28.
* Have screening or prior (in the last 12 months) amyloid PET imaging demonstrating amyloid binding based on qualitative analysis (visual read). Amyloid PET imaging results will be shared with participants, and scans may be used by participants for future research use.
* A brain MRI that supports a diagnosis of AD, with no evidence of significant neurologic pathology.
* Medications taken for symptomatic treatment of AD must be maintained on a stable dosage regimen for at least 30 days before screening visit.
* The subject has an appropriate caregiver capable of accompanying subject on all visits.
* Signed and dated written informed consent obtained from the subject and the subject's legally authorized representative or caregiver (if applicable).

Inclusion criteria for subjects with a diagnosis of Progressive Supranuclear Palsy (PSP)

* Males and females aged 50 to 90 years.
* Has a clinical diagnosis of probable PSP based on the NINDS and Society for PSP (NINDS-PSP) criteria (Litvan, et al 1996).
* Have screening or prior DaTscan SPECT imaging demonstrating evidence of dopamine transporter deficit based on visual read.
* A brain MRI that supports a diagnosis of PSP, with no other evidence of significant neurologic pathology
* Medications taken for symptomatic treatment of PSP must be maintained on a stable dosage regimen for at least 30 days before screening visit.
* The subject has an appropriate caregiver capable of accompanying subject, if necessary.
* Signed and dated written informed consent obtained from the subject and the subject's legally authorized representative or caregiver (if applicable).

Exclusion Criteria:

* Exclusion Criteria (for All subjects)

  * Current or prior history (in the last 12 months) of any alcohol or drug abuse.
  * Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
  * Subject has received an investigational drug or device within 30 days of screening
  * Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 mSv, which would be above the acceptable annual limit established by the US Federal Guidelines.
  * Pregnancy, lactating or breastfeeding.
  * Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Unsuitable veins for repeated venipuncture.
  * MRI exclusion criteria include: Findings that may be responsible for the neurologic status of the patient such as significant evidence of cerebrovascular disease (more than two lacunar infarcts, any territorial infarct >1cm3, or deep white matter abnormality corresponding to an overall Fazekas scale of 3 with at least one confluent hyperintense lesion on the FLAIR sequence that is ≥20 mm in any dimension), infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with CNS disease.
  * Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.

Exclusion criteria for subjects with AD:

• Has received treatment that targeted Aβ or tau within the last 3 months.

Exclusion criteria for subjects PSP:

* Ongoing treatment with methylphenidate, modafinil, metoclopramide, alpha methyldopa, reserpine, or amphetamine derivative for subjects requiring DaTscan imaging.
* Subjects may take stable doses of bupropion, however this medication must be held for at least 12 hours prior to DaTscan imaging.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Tracer uptake will be evaluated in regions of interest for analysis of regional [18F]MNI-958 binding/uptake and expressed in SUV by using established methods for normalization for 4 AD, 7 PSP, and 3 HV subjects. | 1 year
  Target regions of interest in the standard volume of interest (VOI) template, will be used for tracer uptake quantitation of potentially increased binding to tau pathology will correspond in particular to the cortical regions of the brain.
  Descriptive statistics will be applied to describe the tau deposition by region as measured by [18F]MNI-958.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, M.D., Ph. D, Principal Investigator — Invicro
Locations (1):
- Invicro, New Haven, Connecticut, United States

REFERENCES:
- See also: Description Related Info — http://www.invicro.com